CLINICAL TRIAL: NCT00294411
Title: Vaginal Birth After Caesarean Section - Effect on Maternal Psychosocial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4423/03M
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Vaginal Birth After Cesarean

INTERVENTIONS:
Procedure: elective cesarean section

SUMMARY:
The incidence of caesarean section has reached 15-20% in most developed countries. Encouraging vaginal birth after caesareans section (VBAC) has been considered a key component of a strategy to reduce the caesarean section rate. Most medical literature has focused on the efficacy of VBAC in reducing the caesarean section rate and the physical safety of successful VBAC. However, 30%-40% of these women fail to achieve a vaginal delivery. Little is known about how the uncertainty of labour outcome and a failed VBAC impact on the psychosocial function of these women. What we do know is that antenatal depression and unplanned caesarean section are major risk factors for postpartum depression, which in turn is the major cause of maternal mortality in many developed countries including Hong Kong. We propose to study a cohort of women with a prior caesarean section and presenting with a subsequent pregnancy for care. After consent and recruitment, these subjects will be randomly assigned to have a repeat caesarean section or VBAC. The medical outcomes, overall satisfaction of the subjects with the care they received, and the short-term psychosocial function of these subjects will be studied. The result of this study will provide important information that would be useful in assisting women to decide the mode of delivery after a prior caesarean section. The Hypothesis is that there is a significant difference in psychosocial function between these 2 groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* women who agree for vaginal birth after prior cesarean section and who had no previous history of vaginal delivery

Exclusion Criteria:

* Inability or unwillingness to give informed consent. Multiple pregnancy, more than one previous caesarean section, and a previous classical caesarean section, presence of other contra-indications to vaginal birth

Min Age: 0 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-12

PRIMARY OUTCOMES:
General Health Questionnaire (GHQ)

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory
Beck Depression Inventory
Edinburgh Postnatal Depression Scale
Client Satisfaction Questionnaire
MRC Social Performance Schedule
WHO Quality of Life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tze Kin LAU, MD, Principal Investigator — Chinese University of Hong Kong